CLINICAL TRIAL: NCT01116934
Title: Observational Study on Cytokine Production by Leukocytes of Papillon-Lefèvre Syndrome Patients and Healthy Probands in Whole Blood Cultures
Brief Title: Cytokines in Papillon-Lefèvre Syndrome
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Peter Eickholz, Prof. Dr. med. dent., Goethe University
Other Study IDs: PLS-Cytokines
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Papillon-Lefevre Disease
Keywords: blood culture, IL-1β, IL-6, IL-8, IP-10, interferon-gamma
MeSH Terms: conditions — Papillon-Lefevre Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PLS patients: Eight PLS patients (one female) from 6 families.
- Healthy controls: Healthy donors had abstained from taking drugs for two weeks prior to the study. Due to wide spread use of oral contraceptives only male probands were chosen.

SUMMARY:
Papillon-Lefèvre syndrome (PLS) is characterised by aggressively progressive periodontitis combined with palmo-plantar hyperkeratosis. It is caused by "loss of function" mutations in the cathepsin C gene. The hypothesis behind this study is that PLS patients' PMNs produce more proinflammatory cytokines to compensate for their reduced capacity to neutralize leukotoxin and to eliminate Aggregatibacter actinomycetemcomitans. Production of more interleukin (IL)-8 would result in the attraction of more PMNs. Thus, the aim of this study was to evaluate the cytokine profile in PLS patients' blood cultures.

DETAILED DESCRIPTION:
MATERIAL AND METHODS Materials Lipopolysaccharide (LPS; Escherichia coli, serotype R515) was purchased from Alexis (Lausen, Switzerland) and adenosine triphosphate (ATP) from Sigma (Deisenhofen, Germany). Tumor necrosis factor α (TNF-α) was kindly provided by the Knoll AG (Ludwigshafen, Germany). IL-1β was from Invitrogen/Biosource (Karlsruhe, Germany).

Patients and healthy donors Five patients with established diagnose of PLS are under periodontal treatment at the Department of Periodontology, Center for Dental, Oral, and Maxillofacial Medicine (Carolinum) of the Johann Wolfgang Goethe-University Frankfurt am Main. Antiinfective therapy with adjunctive antibiotics has been rendered to all of them and they are under regular and frequent supportive therapy. The Department of Periodontology has contact to additional 5 PLS patients that are edentulous or under periodontal therapy elsewhere. All patients underwent complete oral examinations as well as inspection of the skin of the palms and soles. Each adult patient or parents received clinical and genetic counselling, and signed a consent form, approved by the ethic committees of the Universities of Dresden and Frankfurt/Main. Clinical data and mutations of all patients have been reported before. All these patients were invited to take part in this study. Healthy donors had abstained from taking drugs for two weeks prior to the study. Due to wide spread use of oral contraceptives only male probands were chosen. The study complied with the rules of the Declaration of Helsinki and was approved by the Institutional Review Board for Human Studies of the Medical Faculty of the Johann Wolfgang Goethe-University Frankfurt/Main (Application# 31/05). All participating individuals were informed on risks and benefit as well as the procedures of the study and gave written informed consent.

Whole blood culture Heparinized blood was mixed with an equal volume of culture medium (RPMI 1640 supplemented with 25 mM HEPES (2-[4-(2-hydroxyethyl)piperazin-1-yl]ethanesulfonic acid), 100 U/ml penicillin, 100 µg/ml streptomycin) and 1 ml aliquots were transferred into loosely sealed round-bottom polypropylene tubes (Greiner, Germany). Whole blood cultures were kept at 37 oC and 5 % CO2 for the indicated time periods. Thereafter, cell-free plasma/RPMI samples were obtained by centrifugation and stored at -70oC until assessment of cytokine concentrations by enzyme linked immunosorbent essay (ELISA). Experiments were started within 60 min of blood withdrawal. Thus, the whole blood cultures consisted of the whole range of white blood cells as well as erythrocytes. Except for determination of IL-1β release, cultures were either kept as unstimulated control or stimulated with LPS (10 or 100 ng/ml), or with the combination of IL-1β plus TNF-α (50 ng/ml each) for 24h. For determination of IL-1β release, cells were kept as unstimulated control or were stimulated with Toll-like receptor 4 ligand LPS (100 ng/ml) for altogether 5h. For efficient release of IL-1β from activated cultures, LPS was combined with ATP (2 mM) which was added during the last 2h of the 5h stimulation period in order to achieve activation of the purinoreceptor P2X7.

Analysis of cytokine release by ELISA analysis Concentrations of IL-8, IL-6, interferon-inducible protein (IP)-10, interferon (IFN) gamma (Pharmingen/BD Biosciences), and IL-1β, (R&D Systems), in plasma/RPMI samples were determined by ELISA according to the manufacturers' instructions.

Statistics The individual patient or proband was defined as statistical unit. Data are shown as median with interquartile range and are presented as pg/ml (IL-1β, IL-6, IP-10) or as ng/ml (IL-8). Medians were compared between PLS patients and healthy volunteers using the non parametric Mann Whitney U test. Statistical analysis was performed using a computer program (Systat for Windows version 10.0, Systat Inc., Evanston, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of PLS

Exclusion Criteria:

* No written informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 5 patients with established diagnose of PLS are under periodontal treatment at the Department of Periodontology, Center for Dental, Oral, and Maxillofacial Medicine (Carolinum) of the JWG-University Frankfurt am Main. Antiinfective therapy with adjunctive antibiotics has been rendered to all of them and they are under regular and frequent supportive therapy. The Department of Periodontology has contact to additional 5 PLS patients that are edentulous or under periodontal therapy elsewhere.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2006-07; Primary Completion 2007-01 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Eickholz, Prof. Dr., Study Chair — JWG-University
Locations (1):
- Department of Periodontology, Center for Dental, Oral, and Maxillofacial Medicine (Carolinum), JWG-University, Frankfurt am Main, Germany

REFERENCES:
- [Background] Eickholz P, Kugel B, Pohl S, Naher H, Staehle HJ. Combined mechanical and antibiotic periodontal therapy in a case of Papillon-Lefevre syndrome. J Periodontol. 2001 Apr;72(4):542-9. doi: 10.1902/jop.2001.72.4.542. PMID 11338309
- [Background] Noack B, Gorgens H, Hoffmann T, Fanghanel J, Kocher T, Eickholz P, Schackert HK. Novel mutations in the cathepsin C gene in patients with pre-pubertal aggressive periodontitis and Papillon-Lefevre syndrome. J Dent Res. 2004 May;83(5):368-70. doi: 10.1177/154405910408300503. PMID 15111626
- [Background] Lux CJ, Kugel B, Komposch G, Pohl S, Eickholz P. Orthodontic treatment in a patient with Papillon-Lefevre syndrome. J Periodontol. 2005 Apr;76(4):642-50. doi: 10.1902/jop.2005.76.4.642. PMID 15857107
- [Background] Schacher B, Baron F, Ludwig B, Valesky E, Noack B, Eickholz P. Periodontal therapy in siblings with Papillon-Lefevre syndrome and tinea capitis: a report of two cases. J Clin Periodontol. 2006 Nov;33(11):829-36. doi: 10.1111/j.1600-051X.2006.00992.x. Epub 2006 Sep 13. PMID 16970621
- [Background] Noack B, Gorgens H, Schacher B, Puklo M, Eickholz P, Hoffmann T, Schackert HK. Functional Cathepsin C mutations cause different Papillon-Lefevre syndrome phenotypes. J Clin Periodontol. 2008 Apr;35(4):311-6. doi: 10.1111/j.1600-051X.2008.01201.x. Epub 2008 Feb 20. PMID 18294227

RESULTS

PARTICIPANT FLOW:
Groups:
- Papillon-Lefèvre Syndrome (PLS) Patients: 8 PLS patients (one female) from 6 families
- Healthy Controls: 9 healthy donors
Period: Overall Study
Arm/Group | Papillon-Lefèvre Syndrome (PLS) Patients | Healthy Controls
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PLS Patients: 8 PLS patients (one female) from 6 families
- Total: Total of all reporting groups
Arm/Group | PLS Patients | Healthy Controls | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 0 | 5
  Between 18 and 65 years | 3 | 9 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  Germany | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Serum Concentrations of Interleukin (IL)-1 Beta
Description: Concentrations of IL-8, IL-6, IP-10, interferon (IFN)-gamma, and IL-1 beta, in plasma/RPMI samples were determined by enzyme linked immunosorbent assay (ELISA) according to the manufacturers' instructions
Time Frame: 2006
Population: Samples were stimulated with 100 ng/ml lipopolysaccharide (LPS)
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Papillon-Lefèvre Syndrome (PLS) Patients | Healthy Controls
Number analyzed (Participants) | 8 | 9
pg/ml
  interleukin-1 beta | 1100.00 [896.21 to 2572.10] | 896.21 [771.15 to 2014.00]
  interleukin-6 | 65559 [40365 to 108260] | 45734 [34056 to 66365]
  interferon-inducible protein-10 | 12902.5 [8105.5 to 15735.5] | 11563 [9164 to 19758]
  interferon gamma | 3704.5 [2629.5 to 4372.8] | 3317.4 [2538.5 to 5487.8]
  interleukin-8 | 50520 [29280 to 79870] | 44390 [24680 to 46580]

ADVERSE EVENTS:
Time Frame: Patients were asked to report AEs from blood sampling if they occured.
Arm/Group | PLS Patients | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes